CLINICAL TRIAL: NCT00187967
Title: Blood Activation During Cardiopulmonary Bypass Using Roller or Centrifugal Pumps
Brief Title: Cardiopulmonary Bypass (CPB) Pumps and Blood Activation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PHRC 03-03
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2007-09-26 (Estimated); Status verified 2005-09

CONDITIONS: Cardiopulmonary Bypass; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Cardiopulmonary Bypass

INTERVENTIONS:
Device: pumps used for cardiopulmonary bypass

SUMMARY:
Blood activation induced by cardiopulmonary bypass may compromise the postoperative outcome. The goal of this study is to compare blood activation induced by cardiopulmonary bypass performed with centrifugal pump or roller pump in patients undergoing coronary artery surgery.

ELIGIBILITY:
Inclusion Criteria:

* Men undergoing coronary artery bypass grafting using cardiopulmonary bypass
* Aspirin therapy

Exclusion Criteria:

* Redo surgery
* Acute coronary syndrome requiring urgent surgery
* Oral anticoagulant therapy
* Organ dysfunction or chronic inflammatory disease
* Surgery other than coronary artery bypass grafting

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Dates: Start 2005-01

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Baufreton, MD, PhD, Principal Investigator — University Hospital of Angers, France
Locations (1):
- University Hospital of Angers, Angers, France